CLINICAL TRIAL: NCT00036114
Title: Study of Aripiprazole in the Treatment of Patients With Psychosis Associated With Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Purpose: Treatment
Other Study IDs: CN138-004
Record Dates: First submitted 2002-05-07; First posted 2002-05-09 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2011-04

CONDITIONS: Alzheimer Disease
Keywords: Psychosis associated with dementia of the Alzheimer's type
MeSH Terms: conditions — Alzheimer Disease | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
The purpose of this study is to learn if aripiprazole is safe and effective in the treatment of psychosis associated with dementia of the Alzheimer's type.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized patients with Alzheimer's

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Local Institution, Tuscaloosa, Alabama
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Cerritos, California
  - Local Institution, Granada Hills, California
  - Local Institution, Los Angeles, California
  - Local Institution, San Diego, California
  - Local Institution, Torrance, California
  - Local Institution, Denver, Colorado
  - Local Institution, Hamden, Connecticut
  - Local Institution, Miami, Florida
  - Local Institution, North Miami Beach, Florida
  - Local Institution, West Palm Beach, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Augusta, Georgia
  - Local Institution, Macon, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, North Chicago, Illinois
  - Local Institution, Springfield, Illinois
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Newton Center, Massachusetts
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Wellesley Hills, Massachusetts
  - Local Institution, Lyons, New Jersey
  - Local Institution, Albany, New York
  - Local Institution, Lawrence, New York
  - Local Institution, Montrose, New York
  - Local Institution, Northport, New York
  - Local Institution, White Plains, New York
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Beachwood, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Hershey, Pennsylvania
  - Local Institution, Austin, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Wichita Falls, Texas
  - Local Institution, Bennington, Vermont
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Seattle, Washington

REFERENCES:
- [Derived] Muhlbauer V, Mohler R, Dichter MN, Zuidema SU, Kopke S, Luijendijk HJ. Antipsychotics for agitation and psychosis in people with Alzheimer's disease and vascular dementia. Cochrane Database Syst Rev. 2021 Dec 17;12(12):CD013304. doi: 10.1002/14651858.CD013304.pub2. PMID 34918337